CLINICAL TRIAL: NCT05838118
Title: Washed Microbiota Transplantation (WMT) for Chronic Kidney Disease (CKD): a Open Label, Multicenter Trial
Brief Title: Washed Microbiota Transplantation (WMT) for Chronic Kidney Disease (CKD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Hospital of Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FamingZhang
Record Dates: First submitted 2023-04-08; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-01

CONDITIONS: CKD
Keywords: Fecal Microbiota Transplantation (FMT); Chronic Kidney Disease (CKD)
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Fecal Microbiota Transplantation; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Washed Microbiota Transplantation to treat Chronic Kidney Disease (Other)
  Interventions: Drug: Fecal Microbiota Transplantation
- Standard of Care for Chronic Kidney Disease (Other)
  Interventions: Other: Standard of Care for Chronic Kidney Disease

INTERVENTIONS:
Drug: Fecal Microbiota Transplantation — Biologically active human fecal fluid (donor stool) is provided in fluid form.
  Arms: Washed Microbiota Transplantation to treat Chronic Kidney Disease
Other: Standard of Care for Chronic Kidney Disease — Patients accepted oral drug or dialytic therapy like they used to be to treat CKD.
  Arms: Standard of Care for Chronic Kidney Disease

SUMMARY:
Wahsed microbiota transplantation (WMT) is a novel and promising therapeutic method for Chronic Kidney Disease (CKD). This clinical trail aims to evaluate the efficacy and safety of WMT in the treatment of CKD.

DETAILED DESCRIPTION:
Although the therapeutic methods progress, numerous patients with Chronic Kidney Disease (CKD) can not avoid the clinical outcome of end-stage renal disease. CKD still needs novel treatment to significantly improve the survival quality of the patients.

Gut microbiota has been verified to have relation with immunity. Immunity plays a role in many chronic kidney disease, such as IgA nephropathy, membranous nephropathy and so on. Fecal microbiota transplantation (FMT) is a novel, safe, convenient therapeutic treatment which transplant gut microbiota from donor to patient to rebuild a gut microecology.

This study aims to evaluate the efficacy and safety of FMT in CKD patients. Patients in this study will undergo three times WMT. The primary outcome measure was the clinical remission efficacy rate in the CKD patients. The secondary outcome measure was the safety of WMT in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with chronic kidney disease without WMT in the past three months
* Able to tolerate colonoscopy
* Receiving rescue FMT from the China Microbiota Transplantation System
* Suitable and compatible with WMT treatment
* Patients who can fully understand the content of informed consent for this trial and voluntarily sign a written informed consent form
* Able to receive follow-up examinations, follow-up examinations and retain specimens on time

Exclusion Criteria:

* Patients will be excluded from the analysis if they are not followed up for at least 12 weeks post-FMT
* Antibiotics or probiotics within 4 weeks prior to enrollment
* Patients with anxiety, depression, mental or legal disabilities
* Patients with fulminant type, massive bloody stools, and severe illness unable to tolerate colonoscopy
* Other patients deemed unsuitable for enrollment by the investigator

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-20 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Blood Creatinine | 1 week, 4 week, 12 week
  Patients' Laboratory Change from Baseline Blood Creatinine
Changes in 24-hour Urine Protein | 1 week, 4 week, 12 week
  Patients' Laboratory Change from Changes in 24-hour urine protein

OTHER OUTCOMES:
Rate of Adverse Events | 4 week, 12 week following WMT
  The rate of adverse events after Washed microbiota transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated of Nanjing Medical University, Nanjing, Jiangsu, China

REFERENCES:
- [Result] Zhu H, Cao C, Wu Z, Zhang H, Sun Z, Wang M, Xu H, Zhao Z, Wang Y, Pei G, Yang Q, Zhu F, Yang J, Deng X, Hong Y, Li Y, Sun J, Zhu F, Shi M, Qian K, Ye T, Zuo X, Zhao F, Guo J, Xu G, Yao Y, Zeng R. The probiotic L. casei Zhang slows the progression of acute and chronic kidney disease. Cell Metab. 2021 Oct 5;33(10):2091-2093. doi: 10.1016/j.cmet.2021.08.015. No abstract available. PMID 34614411
- [Result] Xu KY, Xia GH, Lu JQ, Chen MX, Zhen X, Wang S, You C, Nie J, Zhou HW, Yin J. Impaired renal function and dysbiosis of gut microbiota contribute to increased trimethylamine-N-oxide in chronic kidney disease patients. Sci Rep. 2017 May 3;7(1):1445. doi: 10.1038/s41598-017-01387-y. PMID 28469156
- [Result] Xu L, Guo J, Moledina DG, Cantley LG. Immune-mediated tubule atrophy promotes acute kidney injury to chronic kidney disease transition. Nat Commun. 2022 Aug 19;13(1):4892. doi: 10.1038/s41467-022-32634-0. PMID 35986026
- [Result] Lu J, Chen PP, Zhang JX, Li XQ, Wang GH, Yuan BY, Huang SJ, Liu XQ, Jiang TT, Wang MY, Liu WT, Ruan XZ, Liu BC, Ma KL. GPR43 deficiency protects against podocyte insulin resistance in diabetic nephropathy through the restoration of AMPKalpha activity. Theranostics. 2021 Mar 4;11(10):4728-4742. doi: 10.7150/thno.56598. eCollection 2021. PMID 33754024